CLINICAL TRIAL: NCT05566743
Title: A Randomized Phase II Study Evaluating Maintenance Therapy After First Line Induction Chemotherapy in Metastatic Cancer Pancreas
Brief Title: A Study Evaluating Maintenance Therapy After First Line Chemotherapy in Metastatic Cancer Pancreas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Nahla Atef Shabaan, assistant lecturer of clinical oncology and nuclear medicine, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 10001
Record Dates: First submitted 2022-09-22; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Cancer of Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the maintenance arm (Experimental): in this arm patients will receive 4 months of induction FOLFRINOX then maintenance capecitabine
  Interventions: Drug: Capecitabine
- the control arm (Other): in this arm patients will receive 4 months of FOLFRINOX then kept under follow-up
  Interventions: Other: follow up

INTERVENTIONS:
Drug: Capecitabine — maintenance capecitabine after 4 months of FOLFRINOX
  Other Names: Xeloda
  Arms: the maintenance arm
Other: follow up — follow up after 4 months of FOLFRINOX
  Arms: the control arm

SUMMARY:
A randomized phase II study evaluating maintenance therapy after first line induction chemotherapy in metastatic cancer pancreas.

DETAILED DESCRIPTION:
In this study, we aim to evaluate the role of maintenance capecitabine by comparing 2 arms of metastatic cancer pancreas patients in the first line , the first arm will receive 4 months of induction FOLFRINOX the maintenance capecitabine and the second arm will receive 4 months of FOLFRINOX then kept under follow-up:

•Primary end point: PFS.

•Secondary end points: OS, QOL and Toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive adenocarcinoma of pancreas.
* Stage 4 disease according to The American Joint Committee on Cancer (AJCC the 8th Edition) 2017.
* Measurable metastases according to RECIST 1.1.
* Patients underwent surgical resection and postoperative evaluation revealed distant metastasis.
* Patients with age ranging from 18 to 69.
* WHO performance status 0-1.
* An adequate bone marrow reserve and adequate liver and renal function as follow: Neutrophils ≥ 1500 cell/dl, Platelets ≥ 100,000 cell/dl, Hemoglobin ≥ 9.0 g/dl, Total bilirubin < 1.5 × upper normal level (UNL), SGOT and SGPT < 3 × UNL, Creatinine < 1.5 × UNL or estimated GFR > 30 ml/min.
* Adjuvant and neoadjuvant chemotherapies will be permitted if administered more than 6 months before inclusion.
* Patients with biliary or gastroduodenal obstruction must have drainage or surgical bypass prior to starting chemotherapy.
* All patients must have signed and dated informed consent form.

Exclusion Criteria:

* Endocrine or acinar pancreatic carcinoma.
* Patients who progressed during FOLFRINOX regimen.
* Pregnancy or breast feeding.
* Patients with complicated systemic diseases such as diabetes, HTN or decompensated liver disease.
* Patients with any serious uncontrolled medical conditions that might compromise study participation: Central nervous system disorders, gastrointestinal tract disorders that interfere with oral medication.
* Patients with history of previous other carcinoma except basal cell carcinoma of the skin, insitu cervical carcinoma or non-metastatic prostate cancer.
* More than grade 1 peripheral neuropathy.
* Brain metastasis.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-11 (Actual); Primary Completion 2023-09-11 (Estimated); Study Completion 2024-09-11 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 months
  that will be calculated from the time of randomization till disease progression or death

SECONDARY OUTCOMES:
OS | 1 year
  that will be calculated from the time of starting of the disease to death (all causes)

CONTACTS AND LOCATIONS:
Overall Officials: Nahla Atef Shabaan, Master, Principal Investigator — Menoufia University
Locations (2):
- Egypt (2):
  - Egypt, Cairo
  - Nahla Atef Shabaan, Cairo

IPD SHARING:
Plan to Share IPD: No